CLINICAL TRIAL: NCT06835790
Title: Comparative 3-year Study of Nissen-sleeve vs. Sleeve Plus Cruroplasty in Obese Patients With Hiatal Hernia
Acronym: HH-N Sleeve
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Collaborators: Clinique saint-Michel de Toulon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-A00367-40
Record Dates: First submitted 2025-02-18; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Hiatal Hernia
MeSH Terms: conditions — Obesity; Hernia, Hiatal | interventions — Hydrogen-Ion Concentration; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nissen sleeve surgery (Experimental)
  Interventions: Diagnostic Test: Ph-measurement; Other: Questionnaires; Diagnostic Test: gastroduodenal transit
- Sleeve plus cruroplasty (Active Comparator)
  Interventions: Diagnostic Test: Ph-measurement; Other: Questionnaires; Diagnostic Test: gastroduodenal transit

INTERVENTIONS:
Diagnostic Test: Ph-measurement — Ph measurement before and after the surgery
Other: Questionnaires — GERD-HRQL Reflux symptom index scale before and after surgery
Diagnostic Test: gastroduodenal transit — Imaging test that uses the properties of X-rays - after the administration of a radiopaque contrast agent (usually barium) - to visualize the upper digestive tract: the esophagus, stomach, and duodenum (the upper segment of the small intestine).

SUMMARY:
The success of laparoscopic sleeve gastrectomy (LSG) is not only due to its proven efficacy in the treatment of obesity and associated to comorbidities in the short and long term, but also because it is considered as less technically complicated compared to other malabsorptive procedures. Unfortunately, the main long-term side effect of LSG appears to be the development of severe gastroesophageal reflux (GERD). This problem is aggravated by the concomitant presence of a hiatal hernia at the time of surgery. Indeed, by causing laxity of the lower esophageal sphincter (LES), the hiatal hernia reduces the barrier functions of the esophageal-gastric junction against the reflux of gastric contents.

The classic combination of sleeve and hiatal hernia treatment by cruroplasty gives contradictory results and several surgeons prefer to perform only the sleeve without addressing the hiatal hernia especially if it is small (<4 cm). For this reason a modification of the usual surgical technique of LSG has been proposed by adding a Nissen fundoplication-Nissen Sleeve (NS). The intentions of this technique were to minimize the rate of postoperative GERD especially for patients with hiatal hernia, to protect the staple line of the angle of His, and finally to provide a safe and effective alternative for patients with a contraindication to LRYGB due to GERD. Although the first results of the technique are encouraging, the realization of the Nissen valve remains a sensitive technical point that can transform a relatively simple procedure like LSG into a more complex procedure like NS. The only test able to directly identify and classify gastric reflux is pH-metry with or without esophageal manometry. Unfortunately, especially due to the difficulty of access to the examination, there are no studies with solid scientific bases that identify the correct conduct to adopt in the case of an obese patient with a hiatal hernia (with or without preoperative reflux).

The main objective of this study is to evaluate the occurence or worsening of GERD at 3 years following a Nissen-sleeve vs. sleeve plus cruroplasty intervention in patients with obesity and hiatal hernia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient,
* Patient with severe obesity (BMI >35) with comorbidity or morbidity (BMI >40),
* Patient awaiting a sleeve gastrectomy,
* Patient with a hiatal hernia <or= 4 cm,
* Patient having undergone a gastroscopy,
* Patient having undergone an esophagogastroduodenal transit (OGDT),
* Patient having been informed and having given their free, informed and written consent,
* Patient affiliated with or beneficiary of a social security scheme.

Exclusion Criteria:

* Patient with poorly controlled diabetes,
* Patient with major esophageal motility disorders,
* Patient with a Hiatal Hernia > 4cm,
* History of bariatric surgery, history of ring,
* Patient refusing pH-metry examination,
* Refusal to participate in the study,
* Patient under legal protection,
* Patient not benefiting from health protection,
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-02 (Estimated); Primary Completion 2028-11-02 (Estimated); Study Completion 2031-11-02 (Estimated)

PRIMARY OUTCOMES:
Appearance of GERD 3 years after surgery. | 3 years
  Occurrence if DeMeester score at 3 years is ≥ 14.72 (<14.72 before surgery) and/or treatment with proton pump inhibitors (PPIs) and/or Reflux Disease Questionnaire score > 10 (≤10 before surgery) and/or GERD-HRQL score > 16 (≤16 before surgery).
Worsening of GERD 3 years after surgery. | 3 years
  Worsening if increase in DeMeester score at 3 years compared to that before the intervention and/or introduction or increase in the dose of PPI compared to that before the intervention and/or increase in the Reflux Disease Questionnaire score at 3 years compared to that before the intervention and/or increase in the GERD-HRQL score at 3 years compared to that before the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint Michel, Toulon, France